CLINICAL TRIAL: NCT05433831
Title: Feasibility of Application of Nutritional Ultrasound in the Diagnosis and Follow-up of Patients With Nutritional Risk at Hospital Discharge: Study on Body Composition and Function: DRECO Study
Brief Title: Application of Nutritional Ultrasound in the Diagnosis and Follow-up of Patients With Nutritional Risk: DRECO Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: K Access Health Projects (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Dr. José Manuel García Almeida, Clinical Management Unit of Endocrinology and Nutrition, Hospital Universitario Virgen de la Victoria
Other Study IDs: ALM-DRECO-2021-01
Record Dates: First submitted 2022-06-16; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Nutrition Disorders; Malnutrition
Keywords: Ultrasonography; Malnutrition; Clinical Nutrition; Disease Related Malnutrition
MeSH Terms: conditions — Nutrition Disorders; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Disease-related malnutrition (DRM) can occur when there is a deficient supply of energy, protein and/or other nutrients, depending on the nutritional needs of each individual at different times of their life cycle or health or disease circumstances. This deficiency induces effects on body composition and tissue and organ function and results in clinical consequences: increased morbidity and mortality associated with different disease processes.

There are techniques for nutritional assessment using assessment tools aimed at morphofunctional diagnosis of malnutrition, in addition to the classical nutritional parameters, such as weight loss, BMI, folds, circumferences, albumin, lymphocytes, cholesterol and intake. New advanced parameters are being incorporated into clinical nutrition and their incorporation into clinical practice is of increasing interest, such as measures derived from bioelectrical impedance (BIA) and phase angle (PhA), dynamometry, functional tests, CRP/prealbumin ratio and muscle ultrasound.

In 2019, the GLIM criteria were published, providing a different vision of how to assess the malnourished patient. Phenotypic criteria include reduction in muscle mass (measured using validated techniques to measure body composition).

The objective of the study is to highlight nutritional ultrasound for measuring muscle and functional status in order to make a more accurate diagnosis and a better prediction of complications and morbidity and mortality in this type of patients.

DETAILED DESCRIPTION:
Prospective, multicenter, uncontrolled clinical study, of routine clinical practice, without drugs or medical devices

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to hospital who in the first week of admission have moderate or high risk of malnutrition according to the MUST and SARC-F screening test using R-MAPP. Appendix
* Patient aged 18 to 85 years.
* Patient who agrees to participate in the study and signs the informed consent.

Exclusion Criteria:

* Hepatic impairment (AST/ALT 3 x upper limit of normal)
* Chronic kidney failure (GFR <45 mL/min)
* Patient with previous ICU stay during the study admission.
* Cancer patients on palliative treatment or ECOG (Eastern Cooperative Oncology Group) ≥ 3.
* Orthopaedic disease that does not allow adequate walking
* Patients with known dementia or others not related to a significant neurological or psychiatric disorder, or any other psychological condition that may interfere with the conduct of the study.
* Patients with eating disorders
* Life expectancy of less than 6 months.
* Patients unable to adequately complete the clinical laboratory assessments required for the study protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age who, in the first week of hospital admission in medical-surgical areas, excluding critical patients, have an assessment of risk of malnutrition according to the MUST/SARC-F (R-MAPP) screening test, will be included.
  If the results show a moderate or high risk of malnutrition, these patients will be invited to participate in the study, and will undergo the morphofunctional assessment, an ultrasound study and the subjective global assessment (SGA).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Nutritional ultrasound measurements: ultrasound with 4-10 cm linear probe. | Patients will be followed over a period of 6 consecutive months
  * Abdominal ultrasound: total, superficial and pre-peritoneal adipose tissue (measured in centimetres).
  * Muscle ultrasound: Area, circumference, axes and adipose tissue (measured in centimetres)

SECONDARY OUTCOMES:
Sociodemographic data: | Patients will be followed over a period of 6 consecutive months
  Age
Sociodemographic data: | Patients will be followed over a period of 6 consecutive months
  Sex
Sociodemographic data: | Patients will be followed over a period of 6 consecutive months
  Educational level
Sociodemographic data: | Patients will be followed over a period of 6 consecutive months
  Toxic habits
Sociodemographic data: | Patients will be followed over a period of 6 consecutive months
  Medical history
Sociodemographic data: | Patients will be followed over a period of 6 consecutive months
  Risk of sarcopenia and moderate to high malnutrition based on MUST and SARC-F screening test using R-MAPP.
Subjective Global Assessment (SGA) | Patients will be followed over a period of 6 consecutive months
  SGA questionnaire. SGA rank indicates the patient's nutritional status according to 3 categories: (1) well nourished, (2) moderate or suspected malnutrition, and (3) severe malnutrition.
Anthropometric data: | Patients will be followed over a period of 6 consecutive months
  Current body weight (measured or estimated)
Anthropometric data: | Patients will be followed over a period of 6 consecutive months
  Usual weight
Anthropometric data: | Patients will be followed over a period of 6 consecutive months
  Adjusted weight (adjusted weight in obese subjects, dry weight without oedema in malnourished subjects)
Anthropometric data: | Patients will be followed over a period of 6 consecutive months
  Height (measured or estimated)
Anthropometric data: | Patients will be followed over a period of 6 consecutive months
  BMI (body mass index)
Anthropometric data: | Patients will be followed over a period of 6 consecutive months
  Arm circumference
Bioelectrical impedance data (model (50 kHz): | Patients will be followed over a period of 6 consecutive months
  TBW (total body water, L),
Bioelectrical impedance data (model (50 kHz): | Patients will be followed over a period of 6 consecutive months
  ECW (extracellular water, L),
Bioelectrical impedance data (model (50 kHz): | Patients will be followed over a period of 6 consecutive months
  ICW (intracellular water, L),
Bioelectrical impedance data (model (50 kHz): | Patients will be followed over a period of 6 consecutive months
  FFM (lean mass, kg),
Bioelectrical impedance data (model (50 kHz): | Patients will be followed over a period of 6 consecutive months
  FM (fat mass, kg),
Bioelectrical impedance data (model (50 kHz): | Patients will be followed over a period of 6 consecutive months
  BCM (body cell mass, kg),
Bioelectrical impedance data (model (50 kHz): | Patients will be followed over a period of 6 consecutive months
  ASMM (appendicular skeletal muscle mass, kg),
Bioelectrical impedance data (model (50 kHz): | Patients will be followed over a period of 6 consecutive months
  SMI (skeletal muscle mass index, kg),
Bioelectrical impedance data (model (50 kHz): | Patients will be followed over a period of 6 consecutive months
  Percent hydration.
Bioelectrical impedance data (model (50 kHz): | Patients will be followed over a period of 6 consecutive months
  % body fat
Blood biochemistry data (at baseline visit, at 3 and 6 months): | Patients will be followed over a period of 6 consecutive months
  albumin
Blood biochemistry data (at baseline visit, at 3 and 6 months): | Patients will be followed over a period of 6 consecutive months
  prealbumin
Blood biochemistry data (at baseline visit, at 3 and 6 months): | Patients will be followed over a period of 6 consecutive months
  C-reactive protein
Blood biochemistry data (at baseline visit, at 3 and 6 months): | Patients will be followed over a period of 6 consecutive months
  total cholesterol
Blood biochemistry data (at baseline visit, at 3 and 6 months): | Patients will be followed over a period of 6 consecutive months
  lymphocytes
Functional parameters: | Patients will be followed over a period of 6 consecutive months
  Timed Up and Go test (TUG): patient sits in a chair and is told to get up (timing starts), walks 3 meters, comes back and sits in the initial chair (timing ends). Interpretation: <20 seconds: normal,> 20 seconds: increased risk of falling.
Functional parameters: | Patients will be followed over a period of 6 consecutive months
  Dynamometry. Three measurements of the dominant hand will be made recording the mean and maximum, measured in kilograms. Jamar® dynamometers are most used in international studies and have several grip positions.
Current patient status: | Patients will be followed over a period of 6 consecutive months
  Hospital stay, mortality at 3 and 6 months, hospital readmissions and complications. The complications occurring and their consequences (resolved/unresolved) must be recorded in the form.
Adherence. | Patients will be followed over a period of 6 consecutive months
  Attendance to study follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: José Manuel García Almeida, PhD, Principal Investigator — Hospital Clínico Virgen de la Victoria, Málaga (España)
Locations (25):
- Spain (25):
  - Servicio de Endocrinología y Nutrición. Complejo Hospitalario Universitario de Ferrol, A Coruña., A Coruña
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Universitario Vall d´Hebron, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario de Cabueñes, Gijón
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario de Jaén, Jaén
  - Complejo Hospitalario Uni. Insular - Materno Infantil, Las Palmas de Gran Canaria
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Clinical Management Unit of Endocrinology and Nutrition. Virgen de la Victoria Clinical Hospital, Málaga, Málaga
  - UGC Endocrinología y Nutrición. Hospital Regional Universitario, Málaga., Málaga
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Servicio de Endocrinología y Nutrición. Hospital Clínico Universitario de Valladolid, Valladolid., Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia Almeida JM, Bellido D, De Luis D, Guzman Rolo G, Olveira G. Protocol for a prospective cohort study on the feasibility of application of nutritional ultrasound in the diagnosis and follow-up of patients with nutritional risk at hospital discharge: study on body composition and function (DRECO). BMJ Open. 2023 Dec 9;13(12):e074945. doi: 10.1136/bmjopen-2023-074945. PMID 38070895